CLINICAL TRIAL: NCT05254613
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study of Subcutaneous ALXN1830 in Healthy Participants
Brief Title: A Study of Single and Multiple SC Doses of ALXN1830 in Healthy Adult Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The justification of the early termination of the trial: the study is early terminated due to the Coronavirus 2019 epidemic.
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: ALXN1830-HV-105; 2019-003496-18 (EudraCT Number)
Record Dates: First submitted 2022-02-15; First posted 2022-02-24 (Actual); Results first posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (7):
- Cohort 1 (Experimental): Participants will receive a single SC dose of ALXN1830 or placebo (750 mg).
  Interventions: Drug: ALXN1830; Drug: Placebo
- Cohort 2 (Experimental): Participants will receive a single SC dose of ALXN1830 or placebo (1500 mg).
  Interventions: Drug: ALXN1830; Drug: Placebo
- Cohort 3 (Experimental): Participants will receive a single SC dose of ALXN1830 or placebo (2250 mg).
  Interventions: Drug: ALXN1830; Drug: Placebo
- Cohort 4 (Experimental): Participants will receive multiple SC doses of ALXN1830 or placebo (300 mg twice weekly; 8 doses total).
  Interventions: Drug: ALXN1830; Drug: Placebo
- Cohort 5 (Experimental): Participants will receive multiple SC doses of ALXN1830 or placebo (750 mg once weekly; 12 doses total).
  Interventions: Drug: ALXN1830; Drug: Placebo
- Cohort 6 (Experimental): Participants will receive multiple SC doses of ALXN1830 or placebo (1500 mg once weekly; 4 doses total).
  Interventions: Drug: ALXN1830; Drug: Placebo
- Cohort 7 (Experimental): Participants will receive multiple SC doses of ALXN1830 or placebo (2250 mg once weekly; 4 doses total).
  Interventions: Drug: ALXN1830; Drug: Placebo

INTERVENTIONS:
Drug: ALXN1830 — ALXN1830 will be administered as SC infusion(s).
Drug: Placebo — Placebo will be administered as SC infusion(s).

SUMMARY:
This study will evaluate the effects of single ascending doses (SAD) and multiple ascending doses (MAD) of ALXN1830 administered subcutaneously (SC) to healthy adult participants.

DETAILED DESCRIPTION:
This Phase 1 study will consist of 3 SAD (Cohorts 1 to 3) and 4 MAD (Cohorts 4 to 7) cohorts. Participants will be randomly assigned in a 6:2 ratio to each of the 7 cohorts to receive either single or multiple doses of ALXN1830 (n = 6 per cohort) or single or multiple doses of placebo (n = 2 per cohort).

ELIGIBILITY:
Inclusion Criteria:

* Satisfactory medical assessment.
* Participants must have had vaccination against pneumococcus (Pneumovax 23 [PPSV23]) at least 28 days, and maximally 4 years prior to Day 1.
* Participants must have had seasonal influenza vaccination for the current season at least 28 days prior to Day 1.
* Body weight within 50 to 90 kg, inclusive, and body mass index (BMI) within the range of 18 to 24.9 kg/m^2, inclusive.
* Must be willing to follow protocol-specified contraception guidance during the study and for up to 3 months after last dose of study drug.

Exclusion Criteria:

* Current/recurrent diseases or relevant medical history.
* Known exposure to therapeutic proteins, such as monoclonal antibodies, including marketed drugs prior to dosing.
* Participants who have prior exposure to ALXN1830.
* Exposure to more than 4 new (small molecule) investigational compounds within 12 months prior to dosing.
* Current enrollment or past participation within the last 90 days before signing of consent in this or any other interventional clinical study.
* Presence of hepatitis B surface antigen (HBsAg) at Screening.
* Positive hepatitis C antibody test result at Screening.
* Positive human immunodeficiency virus (HIV) antibody test at Screening.
* Participants who are either immunocompromised or have one of the following underlying medical conditions: anatomic or functional asplenia (including sickle cell disease); primary antibody deficiencies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2021-01-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217561&parentIdentifier=ALXN1830-HV-105&attachmentIdentifier=2fdd9bd3-253a-4fe0-9698-054f4c776d17&fileName=alxn1830-hv-105-CSR-synopsis_redacted.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217561&parentIdentifier=ALXN1830-HV-105&attachmentIdentifier=46901612-6e50-4247-bb4c-988803b67523&fileName=alxn1830-hv-105-report-body.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217561&parentIdentifier=ALXN1830-HV-105&attachmentIdentifier=f388a320-1ecb-44f3-94bc-ad07ef808b6c&fileName=alxn1830-hv-105-statistical-method_redacted.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217561&parentIdentifier=ALXN1830-HV-105&attachmentIdentifier=ba92f9f8-8d35-40f6-8211-3374cda86a44&fileName=alxn1830-hv-105-protocol-version-3-amendment-2_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to a lack of participant availability caused by the COVID-19 pandemic, the study was terminated on 22 January 2021 after completion of the ALXN1830 subcutaneous 750 milligrams (mg) dose or placebo groups and partial enrollment of the ALXN1830 subcutaneous 1250 mg dose or placebo groups.
Groups:
- ALXN1830 750 mg: Participants received a single dose of ALXN1830 750 mg subcutaneously on Day 1.
- ALXN1830 1250 mg: Participants received a single dose of ALXN1830 1250 mg subcutaneously on Day 1.
- Placebo: Participants received placebo matched to ALXN1830 subcutaneously on Day 1.
Period: Overall Study
Arm/Group | ALXN1830 750 mg | ALXN1830 1250 mg | Placebo
Started | 6 | 3 | 3
Received at Least 1 Dose of Study Drug | 6 | 3 | 3
Completed | 6 | 3 | 2
Not Completed | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety population consisted of all participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | ALXN1830 750 mg | ALXN1830 1250 mg | Placebo | Total
Number analyzed (Participants) | 6 | 3 | 3 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.8 (2.93) | 23.0 (3.46) | 28.3 (5.86) | 24.3 (4.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 1 | 7
  Male | 3 | 0 | 2 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 3 | 3 | 2 | 8
  Race: Chinese | 0 | 0 | 1 | 1
  Race: Other Asian | 1 | 0 | 0 | 1
  Race: Other | 2 | 0 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not of Hispanic, Latino/a, or Spanish Origin | 6 | 3 | 2 | 11
  Another Hispanic, Latino/a, or Spanish Origin | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Secondary Outcome: Area Under The Serum Concentration Versus Time Curve From Time Zero (Dosing) To The Last Quantifiable Concentration (AUC0-t) of ALXN1830
Time Frame: Predose, end of infusion, and 0.5, 2, 4, 8, and 12 hours postdose on Day 1; and Days 2 to 8
Population: The pharmacokinetic (PK) population consisted of all participants who had sufficient serum ALXN1830 concentration data to evaluate PK parameters. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: hour*nanogram/milliliter
Arm/Group | ALXN1830 750 mg | ALXN1830 1250 mg
Number analyzed (Participants) | 1 | 3
hour*nanogram/milliliter | 31.8 | 44.2 (33.7)

2. Secondary Outcome: Percent Change From Baseline in Immunoglobulin G (IgG) Levels at Day 10
Time Frame: Baseline, Day 10
Population: The pharmacodynamic (PD) population consisted of all participants who had sufficient serum IgG data to evaluate pharmacodynamics effects.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ALXN1830 750 mg | ALXN1830 1250 mg | Placebo
Number analyzed (Participants) | 6 | 3 | 3
percent change | -36.137 (3.7163) | -39.044 (2.0933) | -2.369 (6.6831)

3. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibodies (ADA)
Time Frame: Baseline up to Day 64
Population: The immunogenicity population consisted of all participants who had ADA sample collected.
Measure: Count of Participants; unit: Participants
Arm/Group | ALXN1830 750 mg | ALXN1830 1250 mg | Placebo
Number analyzed (Participants) | 6 | 3 | 3
Participants | 4 | 2 | 0

4. Secondary Outcome: Number of Participants With Positive Neutralizing Antibodies (NAbs)
Description: All samples that are confirmed positive for ADA were evaluated for the presence of neutralizing antibodies.
Time Frame: Baseline up to Day 64
Population: The immunogenicity population consisted of all participants who had ADA sample collected. Here, 'Overall number of participants analyzed' = participants with positive ADA.
Measure: Count of Participants; unit: Participants
Arm/Group | ALXN1830 750 mg | ALXN1830 1250 mg | Placebo
Number analyzed (Participants) | 4 | 2 | 0
Participants | 2 | 2 |

5. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: A TEAE was defined as any adverse event (AE) that commences after the start of administration of study drug. An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study drug, whether or not considered related to the study drug. An AE was considered serious if, in the view of the investigator or sponsor, it resulted in any of the following outcomes: death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect. A summary of all serious AEs and other AEs (nonserious) regardless of causality is located in 'Adverse events' Section.
Time Frame: Baseline up to Day 64
Population: The safety population consisted of all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | ALXN1830 750 mg | ALXN1830 1250 mg | Placebo
Number analyzed (Participants) | 6 | 3 | 3
Participants
  AEs | 5 | 3 | 3
  SAEs | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Day 64
Description: The safety population consisted of all participants who received at least 1 dose of study drug.
Arm/Group | ALXN1830 750 mg | ALXN1830 1250 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 5/6 | 3/3 | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALXN1830 750 mg (N=6) | ALXN1830 1250 mg (N=3) | Placebo (N=3)
Viral upper respiratory tract infection (Infections and infestations) | 5 (5) | 3 (3) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (3) | 1 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site discomfort (General disorders) | 0 (0) | 2 (2) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated early due to a lack of participant availability caused by COVID-19 pandemic after completion of the ALXN1830 750 mg dose group and partial enrollment of the ALXN1830 1250 mg dose group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-01-24): https://cdn.clinicaltrials.gov/large-docs/13/NCT05254613/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-24): https://cdn.clinicaltrials.gov/large-docs/13/NCT05254613/SAP_001.pdf